CLINICAL TRIAL: NCT07098442
Title: The Effect of "Standardized and Real Patient Interviews" on Students' Self-Confidence and Self-Efficacy Levels in Nursing Process Education
Acronym: NursingProcess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hilal Gamze Hakbilen, Res. Assist. Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AkdUni
Record Dates: First submitted 2025-07-17; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Nursing Student
Keywords: Nursing Education; Nursing Process; Clinical Education
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study designed as a single-blind randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online Standart Patient (Experimental)
  Interventions: Behavioral: Online Interview Group
- Clinical Real Patient (Experimental)
  Interventions: Behavioral: Clinical Real Patient Group
- Control Group (Active Comparator)
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Control Group — On the first clinical day, students had a 30-45 minute meeting with the patient they were responsible for, which included the instructor.
  Arms: Control Group
Behavioral: Online Interview Group — Before the Interview
  * Preliminary briefings were given by providing a scenario for the standard patient to be interviewed.
  * Students were given the "Interview Guide," "Nursing Process Case Example," and "Tips for Conducting a Successful Interview" documents and were asked to read them before the interview.
  Interview
  • Students conducted a 30-45 minute interview with a pre-determined standard patient.
  After the Interview
  * The instructor, who monitored the interview, debriefed the students.
  * On the first clinical day after the intervention, students conducted a 30-45 minute interview with the patient they were responsible for, which included the instructor.
  Arms: Online Standart Patient
Behavioral: Clinical Real Patient Group — Before the Interview
  * Patients who were willing to be interviewed in the clinic, stable, and physically and psychologically competent were selected, and the faculty member who would monitor the interview provided preliminary information about the interview.
  * Students were provided with the "Interview Guide," "Nursing Process Case Example," and "Tips for Conducting a Successful Interview" documents and were asked to read them before the interview.
  Interview
  • Students conducted a 30-45 minute interview with a real patient in the pre-determined clinic.
  After the Interview
  * The faculty member who monitored the interview debriefed the students.
  * On the first clinical day after the intervention, students had a 30-45 minute interview with the patient for whom they were responsible, which included the faculty member.
  Arms: Clinical Real Patient

SUMMARY:
The research is a single-center, single-blind (participant), pretest-posttest control group randomized controlled study conducted to determine the effect of meeting with a "standard and real patient" on students' self-confidence and self-efficacy levels in the teaching of the nursing process.

DETAILED DESCRIPTION:
The study, designed as a single-blind randomized controlled trial, was conducted with 83 students at Akdeniz University Faculty of Nursing: 27 "online standardized patient," 30 "clinical real patient," and 26 "control group." The Nursing Process topic within the Fundamentals of Nursing course was taught as usual, with 4 hours of theoretical and 8 hours of laboratory practice. One month before the beginning of clinical practice training, students in the "online standardized patient" and "clinical real patient" groups practiced history taking skills with a standardized patient and a pre-selected real patient for 40 minutes. Students in both groups and the control group then practiced interviewing skills at the beginning of the clinical practice training. The effectiveness of the training was measured using the Self-Confidence Scale, the Self-Assessment Form for Learning Experience, and the Interviewing Skills Evaluation Form.

ELIGIBILITY:
Inclusion Criteria:

* No prior experience in clinical practice
* Taking the Fundamentals of Nursing course for the first time,
* Attending the theoretical explanation of the Nursing Process within the Fundamentals of Nursing course and the history-taking skills demonstration given by the instructor.

Exclusion Criteria:

* Refusing to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | It was applied at the first interview with the patient after randomization and immediately after the last interview. (The period between the first interview before going to the clinic and the last interview after clinical application is 3 months).
  General Self-Efficacy Scale: The scale consists of 17 items and three subscales: "initiation," "perseverance," and "effort-persistence." The measurement tool includes 11 reverse-scored items (2, 4, 5, 6, 7, 10, 11, 12, 14, 16, and 17). The total score on the Likert-type scale ranges from 17 to 85. A higher total score indicates a higher self-efficacy belief.
Self confidence | It was applied at the first interview with the patient after randomization and immediately after the last interview. (The period between the first interview before going to the clinic and the last interview after clinical application is 3 months).
  The Self-Confidence Scale was used to determine students' self-confidence levels. The total score obtained from the 33-item, 5-point Likert-type scale ranges from 33 to 165. The individual's self-confidence level is calculated by dividing the total score by the number of items (33). A score below 2.5 indicates low self-confidence, a score between 2.5 and 3.5 indicates moderate self-confidence, and a score above 3.5 indicates high self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing Faculty, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the study has not yet been published in the literature, we do not prefer to share it.

REFERENCES:
- [Background] Wilson RD, Klein JD, Hagler D. Computer-based or human patient simulation-based case analysis: which works better for teaching diagnostic reasoning skills? Nurs Educ Perspect. 2014 Jan-Feb;35(1):14-8. doi: 10.5480/11-515.1. PMID 24716336
- [Background] Olaussen C, Heggdal K, Tvedt CR. Elements in scenario-based simulation associated with nursing students' self-confidence and satisfaction: A cross-sectional study. Nurs Open. 2019 Sep 27;7(1):170-179. doi: 10.1002/nop2.375. eCollection 2020 Jan. PMID 31871700
- [Background] Labrague LJ, McEnroe-Petitte DM, Bowling AM, Nwafor CE, Tsaras K. High-fidelity simulation and nursing students' anxiety and self-confidence: A systematic review. Nurs Forum. 2019 Jul;54(3):358-368. doi: 10.1111/nuf.12337. Epub 2019 Mar 10. PMID 30852844
- [Background] Ozdemir NG, Kaya H. The effectiveness of high-fidelity simulation methods to gain Foley catheterization knowledge, skills, satisfaction and self-confidence among novice nursing students: A randomized controlled trial. Nurse Educ Today. 2023 Nov;130:105952. doi: 10.1016/j.nedt.2023.105952. Epub 2023 Aug 23. PMID 37639878
- [Background] Sarmasoglu S, Dinc L, Elcin M. Using Standardized Patients in Nursing Education: Effects on Students' Psychomotor Skill Development. Nurse Educ. 2016 Mar-Apr;41(2):E1-5. doi: 10.1097/NNE.0000000000000188. PMID 26102639
- [Background] Ordu Y, Caliskan N. The impact of a web-based mind map learning technique on students' nursing knowledge of the nursing process. Int J Nurs Knowl. 2023 Apr;34(2):108-115. doi: 10.1111/2047-3095.12374. Epub 2022 May 20. PMID 35593697
- [Background] Johnson KV, Scott AL, Franks L. Impact of Standardized Patients on First Semester Nursing Students Self-Confidence, Satisfaction, and Communication in a Simulated Clinical Case. SAGE Open Nurs. 2020 Jun 10;6:2377960820930153. doi: 10.1177/2377960820930153. eCollection 2020 Jan-Dec. PMID 33415284
- See also: Akın, A. (2016). Development and Psychometric Properties of Self-Confidence Scale. Abant İzzet Baysal University Journal of Education, 7(2). — https://dergipark.org.tr/tr/download/article-file/16642
- See also: Yıldırım, F., & İlhan, İ. Ö. (2010). Validity and reliability study of the Turkish form of the general self-efficacy scale. Turkish Journal of Psychiatry, 21(4), 301-308. — https://www.turkpsikiyatri.com/PDF/C21S4/301-308.pdf